CLINICAL TRIAL: NCT04721470
Title: Combined Therapy With Conventional Trans-arterial Chemoembolization (cTACE) and Microwave Ablation (MWA) for Hepatocellular Carcinoma >3-<5 cm
Brief Title: Combined Therapy for Hepatocellular Carcinoma >3-<5 cm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohammad Abd Alkhalik Basha, Assistant Professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6615-18-12-2016
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Combined therapy; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Psychotherapy, Multiple

STUDY DESIGN:
Intervention Model Description: Patients were randomized into three groups: 90 underwent TACE (Group 1); 95 underwent MWA (Group 2); and 93 underwent combined therapy (Group 3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined therapy (Experimental): Patients undergoing combined therapy
  Interventions: Procedure: Combined therapy
- Transarterial chemoembolization (Active Comparator): Patients undergoing Transarterial chemoembolization
  Interventions: Procedure: Transarterial chemoembolization
- Microwave ablation (Active Comparator): Patients undergoing Microwave ablation
  Interventions: Procedure: Microwave ablation

INTERVENTIONS:
Procedure: Combined therapy — Patients undergoing combined therapy
  Other Names: Transarterial chemoembolization + Microwave ablation
  Arms: Combined therapy
Procedure: Microwave ablation — Patients undergoing Microwave ablation
  Arms: Microwave ablation
Procedure: Transarterial chemoembolization — Patients undergoing Transarterial chemoembolization
  Arms: Transarterial chemoembolization

SUMMARY:
The purpose of this study is to compare the safety and efficacy of combined therapy with conventional transarterial chemoembolization (cTACE) + microwave ablation (MWA) versus only TACE or MWA for treatment of hepatocellular carcinoma (HCC) >3-<5 cm.

DETAILED DESCRIPTION:
This study aims to compare the safety and efficacy of combined therapy with conventional transarterial chemoembolization (cTACE)+microwave ablation (MWA) versus only TACE or MWA for treatment of hepatocellular carcinoma (HCC) >3-<5 cm.

This randomized controlled trial screened 278 patients with HCC >3-<5 cm. Patients were randomized into three groups: 90 underwent TACE (Group 1); 95 underwent MWA (Group 2); and 93 underwent combined therapy (Group 3). Patients were followed-up with contrast-enhanced CT or MRI. Images were evaluated and compared for treatment response and adverse events based on modified response evaluation criteria in solid tumor. Serum alpha-fetoprotein (AFP) concentration was measured at baseline and during every follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Solitary HCC >3-<5 cm
2. Absence of extra-hepatic metastases
3. Absence of a history of encephalopathy or refractory ascites
4. Child-Pugh class A or B cirrhosis.

Exclusion Criteria:

1. Poor patient compliance
2. Child-Pugh class C cirrhosis
3. Severe coagulation disorders
4. Portal vein thrombosis
5. Renal impairment (6) previous local ablation therapy of HCC

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Adverse events | Up to three years after procedure
  Images were evaluated and compared for adverse events. The adverse events were recorded and classiﬁed following the guidelines of the Society of Interventional Radiology
Treatment Response | One month
  Tumor response was evaluated by CECT or dynamic MRI based on the modified response evaluation criteria in solid tumor (m-RECIST) established by the American Association for the Study of Liver Diseases.
Recurrence rate | 12 months after procedure
  The recurrence rate was measured in relation to management lines.
Overall mortality rate | Three years after procedure
  The mortality rate was measured in relation to management lines.
Progression-free survival | Three years after procedure
  The progression-free survival was measured in relation to management lines.
AFP variation rate | Baseline and 1-2 months after procedure
  The AFP variation rate (ΔAFP) was defined as the percentage of change between the AFP concentration at baseline and the postprocedure AFP concentration after 1-2 months as shown in the following equation:
  ΔAFP (%) = [(AFPbaseline-AFPpostprocedure) /AFPbaseline] ×100%

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad A Basha, Professor, Principal Investigator — Zagazig University, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zaitoun MMA, Elsayed SB, Zaitoun NA, Soliman RK, Elmokadem AH, Farag AA, Amer M, Hendi AM, Mahmoud NEM, Salah El Deen D, Alsowey AM, Shahin S, Basha MAA. Combined therapy with conventional trans-arterial chemoembolization (cTACE) and microwave ablation (MWA) for hepatocellular carcinoma >3-<5 cm. Int J Hyperthermia. 2021;38(1):248-256. doi: 10.1080/02656736.2021.1887941. PMID 33615957